CLINICAL TRIAL: NCT03848286
Title: A Phase 2 Clinical Study To Evaluate the Efficacy and Safety of KL-A167 Injection in Patients With Recurrent or Metastatic Nasopharyngeal Carcinoma (NPC)
Brief Title: KL-A167 Injection in Recurrent or Metastatic Nasopharyngeal Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sichuan Kelun-Biotech Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sichuan Kelun Pharmaceutical Research Institute Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KL167-Ⅱ-05-CTP
Record Dates: First submitted 2019-02-12; First posted 2019-02-20 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2022-03

CONDITIONS: Nasopharyngeal Carcinoma; Recurrent or Metastatic
Keywords: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma; Recurrence; Neoplasm Metastasis | interventions — 18-O-demethylcervinomycin A2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): KL-A167 900 mg intravenously (IV) every-2-weeks (Q2W)
  Interventions: Drug: KL-A167 Injection

INTERVENTIONS:
Drug: KL-A167 Injection — KL-A167 900 mg intravenously (IV) every-2-weeks (Q2W)

SUMMARY:
The study is to evaluate the efficacy of KL-A167 injection in subjects with recurrent/metastatic Nasopharyngeal Carcinoma, as measured by Overall Response Rate (ORR) per the Response Evaluation Criteria in Solid Tumors RECIST Version 1.1

DETAILED DESCRIPTION:
KL167-Ⅱ-05-CTP (NCT03848286) is a single-arm, open-label, multicenter, phase II study of KL-A167 in pts with R/M NPC. Eligible pts were diagnosed with histopathologically confirmed R/M nonkeratinizing NPC and had received ≥ two lines of chemotherapy. Pts received 900 mg KL-A167 every 2 weeks until disease progression, intolerable toxicity, or withdrawal of consent. The primary endpoint was overall response rate (ORR) evaluated by the independent review committee (IRC) according to Response Evaluation Criteria in Solid Tumors Version 1.1.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years old, male or female;
* Subjects with histopathologically confirmed recurrent/metastatic nonkeratinizing differentiated or undifferentiated NPC;
* Subjects with diseases of clinical stage IVB [Staging System of American Joint Committee on Cancer (AJCC) (8th edition)] who have received first line of platinum-containing combination chemotherapy and second line of monotherapy or failure of combination therapy;
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 to 1;
* Expected survival ≥ 12 weeks;
* Subjects with at least one measurable lesion according to RECIST 1.1, and lesions that have been treated with local therapies, such as radiotherapy, cannot be considered as measurable lesions;
* Tissue or tissue samples must be provided for biomarker analysis. Newly obtained tissues are preferred, and archived paraffin slices are acceptable for patients who do not have newly obtained tissues;
* Adequate organ and bone marrow function, as defined below: a) Hematology: neutrophil count (NEUT #) ≥ 1.5 × 10^9/L; platelet count (PLT) ≥ 90 × 10^9/L; hemoglobin concentration ≥ 9 g/dL; b) Hepatic function: aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 × upper limit of normal (ULN); total bilirubin (TBIL) ≤ 1.5 × ULN; ALT and AST ≤ 5 × ULN for subjects with liver metastases; TBIL ≤ 2 × ULN for subjects with liver metastases or Gilbert's syndrome; c) Renal function: creatinine clearance (CCR) ≥ 50 mL/min; d) Coagulation function: international normalized ratio (INR) ≤ 1.5 and activated partial thromboplastin time (APTT) ≤ 1.5 × ULN;
* Subjects who have taken chemotherapeutic drugs which should be discontinued for ≥ 4 weeks before the first dose (mitomycin or nitrosoureas should be discontinued for ≥ 6 weeks); received surgery, molecular targeted therapy, traditional Chinese medicine therapy with anti-tumor indications, radiotherapy, and anti-tumor therapy with immunostimulatory effect which should be discontinued for 4 weeks or more than 5 half-lives; and antibody drugs which should be discontinued for ≥ 12 weeks (≥ 4 weeks after discontinuation of bevacizumab or nimotuzumab is acceptable); moreover, all treatment-emergent adverse events (TEAEs, except for alopecia) should have stabilized and recovered to the level specified in the eligibility criteria or ≤ Grade 1 toxicity (NCI CTCAE V.5.0);
* Subjects of childbearing potential (male or female) must use effective medical contraception during the study and for 6 months after the end of dosing. Women of childbearing potential must have a negative pregnancy test within 72 h before the first dose;
* Subjects voluntarily participate in the study, sign the ICF, and will be able to comply with the protocol-specified visits and relevant procedures.

Exclusion Criteria:

* Subjects with locally advanced disease will not be screened if they can receive radical treatment such as surgery, radical radiotherapy, or radical chemoradiotherapy;
* Metastases to central nervous system;
* History of other malignancies (except for non-melanoma skin cancer in situ, superficial bladder cancer, cervical cancer in situ, gastrointestinal intramucosal cancer, breast cancer, localized prostate cancer that have been cured and have not recurred within 5 years, which are considered acceptable for enrollment by the investigator);
* History of severe allergic diseases, history of serious drug allergy, and known allergy to macromolecular protein preparations or any component of the KL-A167 Injection formulation;
* Prior treatment with anti-PD-1 antibody, anti-PD-L1 antibody, anti-PD-L2 antibody, anti-CTLA-4 antibody, or CAR-T cells (or any other antibody acting on T-cell co-stimulation or checkpoint pathway);
* Palliative radiotherapy (except for bone metastases) scheduled for symptom control during the study;
* Other systemic anti-tumor therapies that may be received during the study;
* Prior anti-tumor vaccine within 3 months prior to the first dose;
* Allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation or autologous hematopoietic stem cell transplantation within 3 months prior to the first dose;
* Active infection, or unexplained fever before the first dose;
* Systemic use of antibiotics within 1 week prior to signing the ICF;
* Any active autoimmune disease or history of autoimmune disease, including, but not limited to, immune-related neurological disorders, multiple sclerosis, autoimmune (demyelinating) neuropathy, Guillain-Barre syndrome, myasthenia gravis, systemic lupus erythematosus (SLE), connective tissue disorder, scleroderma, inflammatory bowel diseases including Crohn's disease and ulcerative colitis, autoimmune hepatitis, toxic epidermal necrolysis (TEN), or Stevens-Johnson syndrome;
* Subjects with hyperthyroidism and organic thyroid disease will not be screened, but those with hypothyroidism treated with a stable dose of thyroid hormone replacement therapy can be enrolled;
* Systemic treatment with steroids (at a dose equivalent to prednisone > 10 mg/day) or other immunosuppressants within 14 days prior to the first dose; Note: Adrenaline replacement therapy at doses equivalent to prednisone ≤ 10 mg/day is allowed for subjects without active immune disease. Topical, intraocular, intra-articular, intranasal, or inhaled corticosteroids (with minimal systemic absorption) are permitted; and short-term use of corticosteroids for prophylaxis (e.g., contrast allergy) or treatment of non-autoimmune conditions (e.g., delayed-type hypersensitivity caused by contact allergens) is permitted.
* Subjects with serious medical conditions, such as cardiovascular disorders like Grade III or higher abnormal cardiac function (NYHA criteria), ischemic heart disease (such as myocardial infarction or angina pectoris), poorly controlled diabetes mellitus (fasting serum glucose ≥ 10 mmol/L), poorly controlled hypertension (systolic blood pressure > 150 mmHg and/or diastolic blood pressure > 100 mmHg), and ejection fraction < 50% by echocardiography;
* QTc interval > 450 msec for males and > 470 msec for females;
* Abnormal ECG findings and additional risks associated with the use of the investigational product in the opinion of the investigator;
* Presence of active hepatitis B (HBV DNA ≥ 2000 IU/mL or 104 copies/mL) or hepatitis C (positive for hepatitis C antibody and HCV RNA above the lower limit of detection of the assay);
* Known history of human immunodeficiency virus (HIV)-positive or known history of acquired immunodeficiency syndrome (AIDS);
* Subjects with known history of interstitial pneumonia, noninfectious pneumonitis, or highly suspicious of interstitial pneumonia; or subjects with conditions that may interfere with the detection or management of suspected drug-related pulmonary toxicity; and asymptomatic subjects with prior drug-induced or radiation noninfectious pneumonitis are allowed to be enrolled;
* Active pulmonary tuberculosis, or previous history of tuberculosis infection but not controlled by treatment;
* Subjects who have received immunotherapy and experienced ≥ Grade 3 immune-related adverse reactions (ADRs);
* Use of any active vaccine against infectious diseases (e.g. influenza vaccine, varicella vaccine, etc.) within 4 weeks prior to the first dose or planned to be used during the study;
* Previous confirmed history of neurological or mental disorders, including epilepsy or dementia;
* History of definite drug abuse or alcohol abuse within 3 months;
* Pregnant or lactating women;
* Participation in other clinical trials within 1 month prior to the first dose;
* Other factors that may affect the efficacy or safety evaluation of this study in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2019-03-06 (Actual); Primary Completion 2021-07-13 (Actual); Study Completion 2022-01-13 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) assess by Independent Review Committee (IRC) | from first patient first visit to 12 month after last patient first dose
  Based on Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1)

SECONDARY OUTCOMES:
ORR assess by investigators | from first patient first visit to 12 month after last patient first dose
  Based on Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1) and Immune-related Response Evaluation Criteria In Solid Tumors 1.1 (irRECIST 1.1)
Progression-Free Survival (PFS) | from first patient first visit to 12 month after last patient first dose
  PFS as measured in accordance with the Response Evaluation Criteria In Solid Tumours (RECIST) version 1.1
Overall Survival (OS) | from first patient first visit to 12 month after last patient first dose
  Overall Survival is defined as the time from registration to death due to any cause, or censored at date last known alive
Disease Control Rate (DCR) | from first patient first visit to 12 month after last patient first dose
  Based on Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1)
Duration of Response (DOR) | from first patient first visit to 12 month after last patient first dose
  Based on Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1)
Time to Response(TTR) | from first patient first visit to 12 month after last patient first dose
  From the date of the first dose of KL-A167 to the time the response criteria are first met

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No